CLINICAL TRIAL: NCT07336563
Title: Development of a Database of Metabolic Cases and Prevalence of Metabolic Liver Dysfunction (MAFLD/MASLD) in Individuals With Metabolic Syndrome Characteristics - Screening Study (ENDOCARE - SCREEN)
Brief Title: ENDOCARE-SCREEN: Metabolic Liver Dysfunction Screening Study
Acronym: ENDOCARE-SCREE
Status: Not yet recruiting | Type: Observational
Sponsor: Jarosław Drobnik (Other)
Responsible Party: Sponsor-Investigator, Jarosław Drobnik, Prof., Endocare, Poland
Organization: Endocare, Poland (Other)
Other Study IDs: ENDOCARE_23/BNBO/2025
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease (MASH) / Nonalcoholic Steatohepatitis (NASH); Metabolic Syndrome; Obesity & Overweight; Obesity Type 2 Diabetes Mellitus; Insulin Resistance Syndrome
Keywords: MASLD; MAFLD; Metabolic syndrome; Liver steatosis; Screening; Ultrasound; Metabolic health
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Syndrome; Obesity; Overweight; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Screening for Metabolic Dysfunction-Associated Steatotic Liver Disease

SUMMARY:
The ENDOCARE-SCREEN study is a single-center, observational, cross-sectional screening study designed to assess the prevalence, phenotypes, and determinants of metabolic dysfunction-associated steatotic liver disease (MASLD/MAFLD) in adults with components of metabolic syndrome. Up to 10,000 participants aged ≥18 years with overweight, obesity, or metabolic risk factors will undergo standardized screening including a health questionnaire, anthropometric measurements, blood pressure assessment, laboratory testing, and liver ultrasound. The study aims to generate a comprehensive metabolic-hepatic dataset integrating clinical, laboratory, imaging, and lifestyle data. Collected data will be used to identify metabolic and behavioral risk factors for MASLD, characterize disease phenotypes, and support the development of predictive models. The ENDOCARE-SCREEN study will also serve as a qualification platform for selecting eligible participants for a subsequent interventional randomized controlled trial (ENDOCARE-SUPPORT). The study involves minimal risk procedures routinely used in clinical practice and follows ethical principles outlined in the Declaration of Helsinki and Good Clinical Practice (GCP) guidelines.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated steatotic liver disease (MASLD/MAFLD) is currently the most common chronic liver disease worldwide and represents the hepatic manifestation of metabolic syndrome. Despite its high prevalence, large-scale standardized screening data integrating metabolic, imaging, and lifestyle factors are limited in Central and Eastern Europe. The ENDOCARE-SCREEN study addresses this gap by implementing a structured screening program in a real-world ambulatory population. The study collects detailed sociodemographic, metabolic, behavioral, and imaging data, allowing for comprehensive phenotyping of liver dysfunction in individuals with metabolic risk. In addition to epidemiological objectives, the study assesses participants' readiness for lifestyle modification and digital health tools, supporting the future implementation of personalized, technology-assisted interventions. Data generated in ENDOCARE-SCREEN will inform clinical decision-making, public health strategies, and the design of subsequent interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years.
* Overweight or obesity (BMI ≥ 25 kg/m²) and/or increased waist circumference and/or at least one metabolic risk factor (e.g., hypertension, dyslipidemia, impaired fasting glucose/prediabetes/type 2 diabetes), as applicable per screening program.
* Participation in the ENDOCARE screening program.
* Ability to provide written informed consent, including consent for processing health-related data

Exclusion Criteria:

* Inability to provide informed consent (e.g., significant cognitive impairment, acute severe psychiatric disorder, language barrier).
* Pregnancy or breastfeeding.
* Known advanced liver diseases at baseline (participants may be excluded from primary analyses and/or described separately, per statistical analysis plan).
* Refusal of key screening procedures (e.g., blood sampling or liver ultrasound) preventing determination of liver status.
* Refusal of data processing under General Data Protection Regulation (GDPR) requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with potential MAFLD/MASLD syndrome
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of MAFLD/MASLD | Baseline (single screening visit)
  Proportion of participants meeting MAFLD/MASLD criteria according to current definitions
Distribution of hepatic steatosis severity on liver ultrasound | Baseline (single screening visit)
  Ultrasound steatosis grade (0-3): mild (1), moderate (2), severe (3).

SECONDARY OUTCOMES:
Association between MAFLD and metabolic syndrome burden | Baseline
  Relationship between MAFLD status and number of metabolic syndrome components
Association between MAFLD and anthropometric parameters | Baseline
  Relationship between MAFLD and body mass index (BMI) and waist circumference
Association between MAFLD and glycemic status | Baseline
  Relationship between MAFLD and diabetes/prediabetes markers (e.g., fasting glucose/HbA1c as collected)
Association between MAFLD and lipid profile | Baseline
  Relationship between MAFLD and lipid parameters as collected in routine labs
Independent predictors of MAFLD and moderate-to-severe steatosis | Baseline
  Multivariable models (e.g., logistic regression) identifying predictors of MAFLD and moderate-to-severe steatosis
Previously undiagnosed MAFLD/liver disease | Baseline
  Proportion of participants with newly identified MAFLD/liver abnormalities during screening
Eligibility yield for the interventional stage | Baseline
  Proportion of screened participants meeting pre-defined qualification criteria for the second stage (ENDOCARE-SUPPORT)

OTHER OUTCOMES:
Behavioral and motivational profiles related to MAFLD | Baseline
  Lifestyle clusters (diet, physical activity, stimulants) in relation to MAFLD presence
Awareness of fatty liver and readiness to change lifestyle | Baseline
  Self-reported awareness of fatty liver disease and readiness to change lifestyle assessed using a structured study-specific ENDOCARE Lifestyle Awareness and Readiness Questionnaire (score 0-10: higher scores indicate greater awareness of fatty liver disease and higher readiness to implement lifestyle changes)
Acceptance and needs regarding digital health/app features | Baseline
  Self-reported preferences to inform ENDOCARE app development

CONTACTS AND LOCATIONS:
Overall Officials: Jarosław Drobnik, Prof. MD, PhD, Principal Investigator — ENDOCARE Medical Center in Wroclaw, POLAND
Locations (1):
- ENDOCARE, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly. De-identified aggregated results may be shared in scientific publications and conference presentations.

REFERENCES:
- See also: Related Info — https://comipowieszbrzuchu.endocare.wroclaw.pl/